CLINICAL TRIAL: NCT04941599
Title: 2-Hydroxybenzylamine (2-HOBA) to Reduce HDL Modification and Improve HDL Function in Familial Hypercholesterolemia (FH)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, MacRae F. Linton, MD, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201575; 2P01HL116263-06 (NIH)
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial Hypercholesterolemia; HDL; LDL; 2-HOBA; HDL Function
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to treatment with either 2-Hydroxybenzylamine (2-HOBA) , a naturally occuring dicarbonyl scavenger, or placebo for 6 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-Hydroxybenzylamine (2-HOBA) (Active Comparator): 2-Hydroxybenzylamine (2-HOBA) 250 mg three tabs TID (po) for 6 weeks.
  Interventions: Drug: 2-Hydroxybenzylamine
- Placebo (Placebo Comparator): Placebo- three tabs TID (po) for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2-Hydroxybenzylamine — 2-Hydroxybenzylamine (2-HOBA) 250 mg three tabs TID (po) for 6 weeks.
  Other Names: 2-HOBA
  Arms: 2-Hydroxybenzylamine (2-HOBA)
Other: Placebo — Placebo 250 mg three tabs TID (po) for 6 weeks.
  Arms: Placebo

SUMMARY:
The Investigators will test the hypothesis that 2-HOBA will reduce modification of HDL and LDL and improve HDL function in humans with heterozygous FH. The Investigators plan to first study subjects with Familial Hypercholesterolemia (FH), treating them with 750 mg of 2-HOBA or placebo every 8 hours for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with heterozygous Familial Hypercholesterolemia.

Exclusion Criteria:

* Myocardial infarction or stroke within the last 6 months
* unstable angina, symptoms of angina within the last 3 months
* NYHA class III or IV heart failure or LVEF < 30%
* poorly controlled hypertension: SBP > 180 mm Hg or DBP > 110 mm Hg,
* pregnancy,
* evidence of a previous acute coronary syndrome,
* current smokers,
* individuals with Type 2 Diabetes Mellitus, obesity (BMI > 30),
* hypertriglyceridemia (fasting TG > 250 mg/dl),
* renal insufficiency (Cr > 1.8),
* hepatic disease (aspartate aminotransferase(AST) or alanine aminotransferase (ALT) > 2x ULN),
* hypothyroidism,
* nephrotic syndrome,
* rheumatoid arthritis,
* systemic lupus erythematosus,
* AIDS or HIV
* history of malignancy of any organ in last 5 years.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-HOBA increases HDL cholesterol efflux capacity. | Baseline to week 6
  Change in HDL cholesterol efflux capacity will be measured by macrophage cholesterol efflux assay.

SECONDARY OUTCOMES:
2-HOBA reduces modification of HDL by Isolevuglandin (Iso-LG). | Baseline to week 6
  Measurement of the Iso-LG-lysine lactam by mass spectrometry.
2-HOBA reduces modification of HDL by malondialdehyde (MDA). | Baseline to week 6
  Measurement of dilysyl-MDA cross-links by mass spectrometry.

OTHER OUTCOMES:
Change in HDL anti-inflammatory function in an in vitro assay of macrophage cytokine production (IL-1B, TNFa, IL-6). | Baseline to week 6
  Measurement of changes in LPS-stimulated macrophage cytokine production(IL-1B, TNFa, IL-6).
Change in HDL anti-oxidant function in an in vitro assay of macrophage reactive oxygen species production. | Baseline to week 6
  Measurement of changes in H2O2-stimulated macrophage reactive oxygen species
Change in HDL microRNA and small noncoding ribonucleic acid (sRNA) composition | Baseline to week 6
  HDL microRNA and sRNA will be measured through high-throughput sequencing with quantitative polymerase chain reaction (qPCR) validation.
Effects of 2-HOBA on HDL and LDL subpopulation sizes | Baseline to week 6
  HDL and LDL subpopulation sizes and particle numbers will be measured by NMR

CONTACTS AND LOCATIONS:
Overall Officials: MacRae F. Linton, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.